CLINICAL TRIAL: NCT06535620
Title: Comparison of the Effect of Red Wine With Alcohol on Flow-mediated Dilation Versus Red Wine Without Alcohol - a Randomized Clinical Trial
Brief Title: Comparison of the Effect of Red Wine With Alcohol on Flow-mediated Dilation Versus Red Wine Without Alcohol
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Cardiologia de Santa Catarina (Other)
Collaborators: Universidade do Sul de Santa Catarina (Other Government)
Responsible Party: Principal Investigator, Daniel Medeiros Moreira, Professor of Cardiology, Instituto de Cardiologia de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 78483823.4.0000.0261
Record Dates: First submitted 2024-07-28; First posted 2024-08-02 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Healthy Diet
Keywords: wine; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- red wine with alcohol (Experimental): The red wine group
  Interventions: Other: red wine with alcohol
- red wine without alcohol (Placebo Comparator): The non-alcoholic wine group
  Interventions: Other: red wine without alcohol

INTERVENTIONS:
Other: red wine with alcohol — 200 ml of red wine - Demi sec Bordeaux wine 'La Dorni' (alcohol content at 20ºC of 10.1% - Alves & Martins Bebidas Especiais LTDA - Bandeirantes, Parana - Brazil)
  Arms: red wine with alcohol
Other: red wine without alcohol — 200 ml of red wine without alcohol - Demi sec Bordeaux wine 'Casa Navaronne' (alcohol content at 20ºC of 0.23% - Alves & Martins Bebidas Especiais LTDA - Bandeirantes, Parana - Brazil)
  Arms: red wine without alcohol

SUMMARY:
Introduction: Cardiovascular diseases (CVDs) are the leading cause of global mortality, despite being preventable. Moderate wine consumption has been associated with one of the preventative approaches due to its benefits on cardiovascular health, including endothelial protection and antioxidant effects, attributed to its chemical composition, such as flavonoids.

Objective: To assess endothelial function through flow-mediated dilation after the consumption of red wine compared to non-alcoholic wine.

Methodology: A parallel, randomized, placebo-controlled clinical trial with a blinded evaluator will be conducted with 20 healthy participants, evaluated at two distinct time points. Participants will be selected to receive either red wine or non-alcoholic wine and will be crossed over after 7 days to receive the opposite beverage from the initial one. The primary outcome will be the change in flow-mediated dilation of the brachial artery pre- and post-intervention in both groups. The secondary outcomes will include the flow-mediated dilation values, brachial artery diameter after the intervention, and measurements of systolic blood pressure (SBP) and diastolic blood pressure (DBP).

ELIGIBILITY:
Inclusion Criteria:

* consume alcohol sporadically

Exclusion Criteria:

* continuous medication, including anti-inflammatories
* pregnant women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-13 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated dilation | 40 minutes after the substance intake
  Evaluate flow-mediated dilation after the consumption of red wine compared to placebo

SECONDARY OUTCOMES:
Heart rate | 40 minutes after the substance intake
  Analyze the difference in heart rate (in bpm) after the consumption of red wine compared to the consumption of non-alcoholic wine.
Blood pressure | 40 minutes after the substance intake
  Analyze the difference in blood pressure (in mmHg) after the consumption of red wine compared to the consumption of non-alcoholic wine.
Brachial artery diameter at rest | 40 minutes after the substance intake
  Evaluate the difference in the diameter (at rest) of the brachial artery (measured in millimeters) before and after consuming red wine.
Brachial artery diameter after endothelial stress | 40 minutes after the substance intake
  Evaluate the difference in the diameter (after endothelial stress) of the brachial artery (measured in millimeters) before and after consuming red wine.

IPD SHARING:
Plan to Share IPD: No